## TREATMENT OF PERI-IMPLANT MUCOSITIS USING AN ER: YAG LASER OR AN ULTRASONIC DEVICE. A RANDOMIZED CLINICAL TRIAL.

Statistical analysis plan NCT 05772299



Statistical analysis plan in the study. "Treatment of periimplant mucositis using an Er: Yag laser or an ultrasonic device. A randomized clinical trial."

The power analysis was based on: If bleeding on probing (BOP) is reduced with  $30\% \pm 10$  in the test group and with a  $30\% \pm 10$  decrease in the control group, detected at alpha= 0.05 and a power of beta= 0.2. The power analysis showed a minimum of 38 individuals to reach a significant difference. It will be foreseen to incorporate 45 individuals if some of the individuals will not fulfil the study.

The IBM SPSS version 28.0 statistical software package (SPSS Inc., Armonk, NY, USA) for personal computer will be used in the statistical analyses.

Statistics will be calculated as means and standard deviation (SD). To compare inter and intra group differences independent t-test (equal variance not assumed), paired t-test and one-way ANOVA test will be used.

For categorical variables non-parametric chi-square test will be used. Statistical significance will be set with 80% and at p< 0.05.

Non visits will be recorded as missing data in the statistics.